CLINICAL TRIAL: NCT06458764
Title: SEXCHECK - Sexual Dysfunction Check-up in Premenopausal Breast Cancer Survivors Taking Endocrine Therapy: A Cross-Sectional Study
Brief Title: Sexual Dysfunction Check-up in Premenopausal Breast Cancer Survivors Taking Endocrine Therapy: A Cross-Sectional Study
Acronym: SEXCHECK
Status: Recruiting | Type: Observational
Sponsor: Candiolo Cancer Institute - IRCCS (Other)
Responsible Party: Principal Investigator, Giada Pozzi, MD, Candiolo Cancer Institute - IRCCS
Other Study IDs: 71/2023
Record Dates: First submitted 2024-06-06; First posted 2024-06-14 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2024-06

CONDITIONS: Breast Cancer Female; Sexual Dysfunction; Premenopausal Breast Cancer
MeSH Terms: conditions — Sexual Dysfunction, Physiological | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Month
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Patients
  Interventions: Other: Questionnaire
- Controls
  Interventions: Other: Questionnaire

INTERVENTIONS:
Other: Questionnaire — none, it's a incidence-prevalence study

SUMMARY:
Primary objectives:

* To estimate Sexual Dysfunction (SD) incidence in premenopausal breast cancer patients treated by surgery and taking endocrine therapy.
* To detect the presence of SD-related distress in the population, as a determining factor in the maintenance of a good quality of life.

Secondary objectives:

* To describe SD characteristics determining the most frequently reported symptoms and correlations with type of surgery or therapeutic regimens.
* Collect baseline data for subsequent randomized trials involving practical interventions with the aim to reduce SD prevalence in this population.

ELIGIBILITY:
Inclusion Criteria:

* women aged ≥18 and ≤ 55
* who underwent surgery for early stage breast cancer
* taking endocrine therapy for at least 3 months
* providing an informed consent and completing the study questionnaires.

Exclusion Criteria:

* withdrawal of the informed consent, at any time

Ages: 18 Years to 55 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Women aged ≥18 and ≤ 55 who underwent surgery for early stage breast cancer, taking endocrine therapy for at least 3 months
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-01 (Estimated)

PRIMARY OUTCOMES:
Sexual Dysfunction (SD) incidence | 6 months
  To estimate Sexual Dysfunction (SD) incidence (physiological parameter) in premenopausal breast cancer patients treated by surgery and taking endocrine therapy.
SD-related distress | 6 months
  To detect the presence of SD-related distress (physiological parameter) in the population, as a determining factor in the maintenance of a good quality of life.

SECONDARY OUTCOMES:
SD characteristics | 6 months
  To describe SD characteristics determining the most frequently reported symptoms and correlations with type of surgery or therapeutic regimens.
Collect baseline data | 6 months
  Collect baseline data for subsequent randomized trials involving practical interventions with the aim to reduce SD prevalence in this population.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Candiolo Cancer Center, Torino, TO, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] McCool ME, Zuelke A, Theurich MA, Knuettel H, Ricci C, Apfelbacher C. Prevalence of Female Sexual Dysfunction Among Premenopausal Women: A Systematic Review and Meta-Analysis of Observational Studies. Sex Med Rev. 2016 Jul;4(3):197-212. doi: 10.1016/j.sxmr.2016.03.002. Epub 2016 Apr 19. PMID 27871953
- [Background] Jing L, Zhang C, Li W, Jin F, Wang A. Incidence and severity of sexual dysfunction among women with breast cancer: a meta-analysis based on female sexual function index. Support Care Cancer. 2019 Apr;27(4):1171-1180. doi: 10.1007/s00520-019-04667-7. Epub 2019 Feb 2. PMID 30712099
- [Background] Seav SM, Dominick SA, Stepanyuk B, Gorman JR, Chingos DT, Ehren JL, Krychman ML, Su HI. Management of sexual dysfunction in breast cancer survivors: a systematic review. Womens Midlife Health. 2015 Nov 2;1:9. doi: 10.1186/s40695-015-0009-4. eCollection 2015. PMID 30766696
- [Background] Du H, Chen C, Yuan F, Hu A, Han J. Correlation analysis of body image level and female sexual dysfunction in young patients with postoperative breast cancer. J Cancer Res Ther. 2022 Sep;18(5):1360-1371. doi: 10.4103/jcrt.jcrt_629_21. PMID 36204884
- [Background] Carmen A, Anne O, Monika S, Daniel E, Johannes G, Verena M, Michael H, Christine B. Does the toxicity of endocrine therapy persist into long-term survivorship?: Patient-reported outcome results from a follow-up study beyond a 10-year-survival. Breast Cancer Res Treat. 2023 Apr;198(3):475-485. doi: 10.1007/s10549-022-06808-9. Epub 2022 Nov 23. PMID 36418518
- [Background] Sousa Rodrigues Guedes T, Barbosa Otoni Goncalves Guedes M, de Castro Santana R, Costa da Silva JF, Almeida Gomes Dantas A, Ochandorena-Acha M, Terradas-Monllor M, Jerez-Roig J, Bezerra de Souza DL. Sexual Dysfunction in Women with Cancer: A Systematic Review of Longitudinal Studies. Int J Environ Res Public Health. 2022 Sep 21;19(19):11921. doi: 10.3390/ijerph191911921. PMID 36231221
- [Background] Qi A, Li Y, Sun H, Jiao H, Liu Y, Chen Y. Incidence and risk factors of sexual dysfunction in young breast cancer survivors. Ann Palliat Med. 2021 Apr;10(4):4428-4434. doi: 10.21037/apm-21-352. PMID 33966393
- [Background] Taylor CE, Meisel JL. Management of Breast Cancer Therapy-Related Sexual Dysfunction. Oncology (Williston Park). 2017 Oct 15;31(10):726-9. PMID 29083465
- [Background] Gorman JR, Lyons KS, Harvey SM, Acquati C, Salsman JM, Kashy DA, Drizin JH, Smith E, Flexner LM, Hayes-Lattin B, Reese JB. Opening the Conversation: study protocol for a Phase III trial to evaluate a couple-based intervention to reduce reproductive and sexual distress among young adult breast and gynecologic cancer survivor couples. Trials. 2022 Sep 2;23(1):730. doi: 10.1186/s13063-022-06665-3. PMID 36056413
- [Background] Advani P, Brewster AM, Baum GP, Schover LR. A pilot randomized trial to prevent sexual dysfunction in postmenopausal breast cancer survivors starting adjuvant aromatase inhibitor therapy. J Cancer Surviv. 2017 Aug;11(4):477-485. doi: 10.1007/s11764-017-0606-3. Epub 2017 Feb 22. PMID 28229275
- [Background] Ljungman L, Ahlgren J, Petersson LM, Flynn KE, Weinfurt K, Gorman JR, Wettergren L, Lampic C. Sexual dysfunction and reproductive concerns in young women with breast cancer: Type, prevalence, and predictors of problems. Psychooncology. 2018 Dec;27(12):2770-2777. doi: 10.1002/pon.4886. Epub 2018 Sep 27. PMID 30203884
- [Background] Maiorino MI, Chiodini P, Bellastella G, Giugliano D, Esposito K. Sexual dysfunction in women with cancer: a systematic review with meta-analysis of studies using the Female Sexual Function Index. Endocrine. 2016 Nov;54(2):329-341. doi: 10.1007/s12020-015-0812-6. Epub 2015 Dec 7. PMID 26643312
- [Background] Fogh M, Hojgaard A, Rotbol CB, Jensen AB. The majority of Danish breast cancer survivors on adjuvant endocrine therapy have clinically relevant sexual dysfunction: a cross-sectional study. Acta Oncol. 2021 Jan;60(1):61-68. doi: 10.1080/0284186X.2020.1813326. Epub 2020 Sep 1. PMID 32869712
- [Background] Gandhi C, Butler E, Pesek S, Kwait R, Edmonson D, Raker C, Clark MA, Stuckey A, Gass J. Sexual Dysfunction in Breast Cancer Survivors: Is it Surgical Modality or Adjuvant Therapy? Am J Clin Oncol. 2019 Jun;42(6):500-506. doi: 10.1097/COC.0000000000000552. PMID 31094713
- [Background] Cobo-Cuenca AI, Martin-Espinosa NM, Sampietro-Crespo A, Rodriguez-Borrego MA, Carmona-Torres JM. Sexual dysfunction in Spanish women with breast cancer. PLoS One. 2018 Aug 31;13(8):e0203151. doi: 10.1371/journal.pone.0203151. eCollection 2018. PMID 30169506
- [Background] Carpenter JS, Reed SD, Guthrie KA, Larson JC, Newton KM, Lau RJ, Learman LA, Shifren JL. Using an FSDS-R Item to Screen for Sexually Related Distress: A MsFLASH Analysis. Sex Med. 2015 Mar;3(1):7-13. doi: 10.1002/sm2.53. PMID 25844170